CLINICAL TRIAL: NCT03864484
Title: An iPad Application-based Intervention for Improving Post-stroke Depression Symptoms: A Pilot Randomized Controlled Trial
Brief Title: iPad Application-based Intervention for Post-stroke Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kibi International University (Other)
Responsible Party: Principal Investigator, Kazuki Hirao, PhD, OT, Assistant Professor, Kibi International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H30-038
Record Dates: First submitted 2019-03-02; First posted 2019-03-06 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Post-stroke Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPad Application + Usual Rehabilitation (Experimental): The experimental group receives usual rehabilitation. In addition, participants watch a video using the iPad Application displaying positive word stimuli.
  Interventions: Device: iPad Application + Usual Rehabilitation
- Usual rehabilitation (Active Comparator): The control group receives usual rehabilitation.
  Interventions: Behavioral: Usual rehabilitation

INTERVENTIONS:
Device: iPad Application + Usual Rehabilitation — The experimental group receives usual rehabilitation. In addition, the experimental group will watch movies using the iPad application for 3 minutes, once daily for 5 weeks.
  Arms: iPad Application + Usual Rehabilitation
Behavioral: Usual rehabilitation — The control group receives usual rehabilitation.
  Arms: Usual rehabilitation

SUMMARY:
We plan to conduct a randomized controlled trial to examine whether usual rehabilitation plus an iPad application-based intervention improves post-stroke depression symptoms compared to usual rehabilitation alone.

The purpose of this pilot randomized controlled trial is to investigate the feasibility of the final randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 40 years and older
* Males and females
* Center for Epidemiologic Studies Depression Scale score ≥16
* Mini Mental State Examination score ≥ 24
* First stroke
* Native language is Japanese
* Written informed consent prior to participation

Exclusion Criteria:

* Major depressive disorder before onset of stroke
* Bilateral hemiplegia
* Vision or hearing deficits that negatively impact everyday life
* Severe aphasia
* Severe unilateral spatial neglect
* Diagnosis of neurodegenerative disease such as Parkinson's disease or multiple system atrophy
* Current life-threatening severe organ failure, musculoskeletal disorders, or cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Depression severity as measured by the Center for Epidemiologic Studies Depression Scale (CES-D) score. | Change from Baseline CES-D at 5 weeks

SECONDARY OUTCOMES:
Health-related quality of life as measured by the 36-item short-form Medical Outcome Study Questionnaire (SF-36). | Change from Baseline SF-36 at 5 weeks
Activities of daily living as measured by Functional Independence Measure (FIM). | Change from Baseline FIM at 5 weeks
Dynamic standing balance as measured by Functional Reach Test (FRT). | Change from Baseline FRT at 5 weeks
Safety is defined as the proportion of patients who experience an intervention-related adverse event or any adverse event during the study. | The period from the start of the intervention to 5 weeks
  Adverse events, whether or not considered causally related to the study intervention, include death and life-threatening illness or injury requiring prolonged hospitalization or resulting in persistent disability.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuki Hirao, PhD, Principal Investigator — Kibi International University
Locations (1):
- Kurashiki Heisei Hospital, Kurashiki, Okayama-ken, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ejiri H, Uchida H, Tsuchiya K, Fujiwara K, Kikuchi S, Hirao K. Effects of Smartphone-Delivered Positive-Word Stimulation on Depressed Mood in People with Subthreshold Depression: Protocol for a Pilot Randomized Controlled Trial. Neuropsychiatr Dis Treat. 2021 Aug 20;17:2739-2748. doi: 10.2147/NDT.S323126. eCollection 2021. PMID 34456565